CLINICAL TRIAL: NCT07186816
Title: SUPERA: Supporting Peer Interactions to Expand Access to Digital Cognitive Behavioral Therapy for Spanish-speaking in the San Francisco Mission Community
Brief Title: SUpport From PEeRs to Expand Access Study - Community
Acronym: SUPERA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Berkeley (Other)
Collaborators: University of California, Irvine (Other); University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 22-36825
Record Dates: First submitted 2025-08-26; First posted 2025-09-22 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Depression, Anxiety
MeSH Terms: conditions — Depression; Anxiety Disorders

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Peer-Support (Experimental)
  Interventions: Device: Behavioral: Supported dCBT
- Control (Active Comparator)
  Interventions: Device: Behavioral: Unsupported dCBT

INTERVENTIONS:
Device: Behavioral: Supported dCBT — In the supported dCBT condition, each patient will receive complete access to the SilverCloud platform. In addition, patients will be assigned a supporter who will provide regular support based on an established coaching support protocol. Supporters will conduct a brief engagement call (30-40 minutes) to provide an overview of SilverCloud, identify goals, and set expectations, introduce themselves, and orient the participant to the role of the peer supporter. Supporters will then provide weekly check-ins through phone calls or messaging. Participants will be able to communicate with the supporters through the platform through messaging or sharing activities for additional discussion. The major goal of the support is to promote use of the platform.
  Arms: Peer-Support
Device: Behavioral: Unsupported dCBT — Unsupported dCBT provides all features of the SilverCloud platform with the exception of support features (structured interactions with supporter and share features). Patients will be provided complete access to SilverCloud and instructed to use it for 8-weeks. Patients will receive weekly automated messages to encourage engagement.
  Arms: Control

SUMMARY:
Investigators will evaluate the implementation of an evidence-based, Spanish-language, digital, cognitive-behavioral therapy (dCBT) intervention (SilverCloud) in the Mission community for Latino patients with depression and/or anxiety. 213 participants will be enrolled in a one-armed trial comparing self-guided vs. supported dCBT (SilverCloud).

ELIGIBILITY:
Inclusion Criteria:

1. PHQ-9 ≥ 10 or GAD-7 ≥ 8
2. Has access to the Internet via smartphone and/or broadband at home, and basic level of technological literacy or willingness to undergo a brief technology use training
3. ≥18 years of age
4. Preference for receiving medical care in Spanish
5. Not in concurrent psychotherapy
6. If currently taking an antidepressant medication, patient must have been on a stable dose for at least 6 weeks, and have no plans to change the dose. We will permit patients on antidepressants to enter the study, as this will increase generalizability. Antidepressant status will be monitored at each assessment to control for those effects, if necessary.

Exclusion Criteria:

1. Currently receiving psychotherapy, as this treatment will be offered as a frontline treatment for depression and anxiety, however, patients are allowed to be referred to treatment while participating in this study and initiation of treatment will be monitored and considered in analyses
2. Visual, hearing, voice, or motor impairment or illiteracy that would prevent completion of study procedures
3. Diagnosis of a psychotic disorder, bipolar disorder, dissociative disorder, or substance use disorder
4. Severe suicidality (as assessed by expressing suicidal ideation, plan, and intent). Although procedures with back-up plans are in place for patients who develop suicidality (see Human Subjects Section), patients assessed with severe suicidality will be referred to more-intensive treatment resources.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 213 (Estimated)
Dates: Start 2025-08-18 (Actual); Primary Completion 2027-03-01 (Estimated); Study Completion 2027-03-01 (Estimated)

PRIMARY OUTCOMES:
Change in Depression at 8 Weeks | Change from Baseline to Week 8
  The primary outcome of symptoms of depression will be measured with the self-report Patient Health Questionnaire-9 (PHQ-9). The PHQ-9 is a 9-item self-report measure of depression. Scores on this measure range from 0 (Not At All) to 3 (Nearly Every Day).
Change in Anxiety at 8 Weeks | Change from Baseline to Week 8
  The primary outcome of symptoms of depression will be measured with the self-report General Anxiety Disorder-7 (GAD-7). The GAD-7 is a 7-item self-report measure of anxiety. Scores on this measure range from 0 (Not At All) to 3 (Nearly Every Day).

CONTACTS AND LOCATIONS:
Locations (1):
- Zuckerberg San Francisco General, San Francisco, California, United States